CLINICAL TRIAL: NCT05227508
Title: A Double-blind, Placebo Controlled, 12-week Treatment Trial in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: The Effect of BRIZO on Lower Urinary Tract Symptoms (LUTS) Related to Benign Prostatic Hypertrophy (BPH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Se-cure Pharmaceuticals Ltd. (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0615-21-RMC
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: BPH Without Urinary Obstruction and Other Lower Urinary Tract Symptoms (LUTS)

STUDY DESIGN:
Intervention Model Description: * Study arm- min. 80 patients
  * Placebo arm- min. 40 patients
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brizo SC012 (Experimental): A capsule containing 400 mg. SC012 (unique soy extract) TWICE A DAY : MORNING , EVENING.
  Interventions: Dietary Supplement: BRIZO
- PLACEBO (Placebo Comparator): A capsule containing 400 mg OF PLACEBO, TWICE A DAY: MORNING , EVENING.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: BRIZO — A capsule containing 400 mg. SC012 (unique soy extract)
  Arms: Brizo SC012
Other: placebo — Comprecel microcrystalline cellulose
  Arms: PLACEBO

SUMMARY:
A randomized, placebo controlled double-blind, 12-week treatment trial in men with moderate to severe symptoms of benign prostatic hyperplasia. The trail is about to examine the effect of Brizo® on reduction of BPH related symptoms.

DETAILED DESCRIPTION:
1. Males in good general health 50 years of age and older, with symptoms of moderate to severe benign prostatic hyperplasia.
2. 120 patients: Study arm- min. 80 patients Placebo arm- min. 40 patients Final Aim for Stat. Sig.: 75% of recruitment group (90 patients)
3. Duration - 12 weeks with 3 visits: 0,6,12 weeks
4. The following procedures are utilized:

   * Physical exams - visit 1,3.
   * Drugs/food supplement usage questionnaire - visit 1.
   * Product supply Control - visit 1,2.3
   * Clinical laboratory tests : psa, cbc, bun - visit 1,3.
   * Uroflowmetry test visit - visit 1,3.
   * IPSS- International Prostate Symptom Score - questionnaire - visit 1, 3.
   * IIEF questionnaire - visit 1, 3.
5. dosage: 1 capsule twice daily (morning & evening) can be taken with or without food

ELIGIBILITY:
Inclusion Criteria:

Males in good general health at least 50 years of age, with symptoms of moderate to severe benign prostatic hyperplasia

Exclusion Criteria:

* Inability to complete the questionnaire.
* Patients with or suspected of having prostate cancer.
* Patients who have undergone a surgical procedure in the past year and / or who have taken medications or supplements in the past six months to treat BPH.
* Patients treated with drugs for kidney / urinary tract problems.
* Allergy to soy.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Improved index in the IPSS test | 12 weeks
  Improvement by 3 points and with a significance of P< 0.05.

SECONDARY OUTCOMES:
Improve UROFLOWMETRY test | 12 WEEKS
  Improve from personal baseline in UROFLOWMETRY test at Week 12 .

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Shoshani, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center - Clalit Health Services, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No